CLINICAL TRIAL: NCT02122965
Title: The Effect of Medication Review in High-risk Emergency Department Patients: Evaluation of a Quality Improvement Program
Brief Title: The Effect of Medication Review in High-risk Emergency Department Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H11-01815
Record Dates: First submitted 2014-04-15; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Adverse Drug Events; Adverse Drug Reactions; Medication-related Problems
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist-led medication review (Experimental): Pharmacist-led medication review in the ED
  Interventions: Other: Pharmacist-led medication review
- Usual care (No Intervention): Usual care includes nurse-led medication reconciliation.

INTERVENTIONS:
Other: Pharmacist-led medication review — Medication review is a structured, critical examination of a patient's medications with the objective of reaching agreement with the patient about treatment, optimizing the medications' impact, and minimizing the number of medication-related problems and adverse drug events.
  Arms: Pharmacist-led medication review

SUMMARY:
Adverse drug events are unintended and harmful events related to medication use and a leading cause of emergency department visits, unplanned hospital admissions and deaths. In the emergency department, physicians frequently misdiagnose adverse drug events leading to treatment delays. Our objective is to evaluate the effect of pharmacist-led medication review in high-risk emergency department patients on prolonged hospital stay.

This prospective multi-centre, quasi-randomized study is nested within an existing quality improvement program. Triage nurses flag incoming emergency department patients at high-risk for adverse drug events by applying a clinical decision rule consisting of four variables (co-morbid conditions, antibiotic use within 7 days, medication changes within 28 days, and age). Consecutive eligible high-risk patients are enrolled into the medication review study, and systematically allocated to pharmacist-led medication review or usual care. In the intervention group, medication review pharmacists collect best-possible medication histories, review the patient's medications for appropriateness and adverse drug events, and communicate the results of medication review to patients, caregivers and physicians. In the usual care group, physicians refer patients to onsite pharmacists for medication management questions on an as needed basis. Health outcomes are assessed using anonymized data linkage to administrative health databases. The primary outcome is the percent of days spent in hospital during the first 30 days after the index emergency department visit

ELIGIBILITY:
Inclusion Criteria:

Consecutive high-risk patients, aged 19 years or older, presenting to a participating emergency department when a medication review pharmacist is on duty are eligible for enrolment.

Exclusion Criteria:

We will exclude patients categorized as Canadian Triage Acuity Score (CTAS) 1 as they require immediate resuscitation, those presenting for multisystem trauma (e.g., penetrating trauma), scheduled visits (e.g., for intravenous antibiotics), sexual assaults, pregnancy-related complications, social problems, and those for whom we cannot link data to administrative records (e.g., out-of-province patients).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10805 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Proportion of days spent in hospital over 30 days | 30 days
  The primary outcome will be the proportion of days spent in hospital during the follow up period. This outcome captures all days in hospital that were incurred during the index admission as well as during any readmissions.

SECONDARY OUTCOMES:
Hospital admission | on the 1 day of medication review
Prolonged hospital stay | 30 days
  Prolonged hospital stay will be defined as a length of stay that is greater than the median length of stay observed by high-risk patents during the pilot period.
Unplanned emergency department re-visit | 7 days
Mortality | 30 days
Unplanned readmission | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Corinne M Hohl, MD, MHSc, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Richmond Hospital, Richmond, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia